CLINICAL TRIAL: NCT01620697
Title: Value of Perirenal Fat Surface as a Risk Factor for Morbidity After Elective Colorectal Surgery
Brief Title: Visceral Obesity and Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Francesco Volonté, MD, MD, University Hospital, Geneva
Other Study IDs: FAT-40-GVA
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Visceral Obesity; Colorectal Surgery; Risk Factor
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Perirenal fat
  Interventions: Procedure: Colorectal surgery

INTERVENTIONS:
Procedure: Colorectal surgery — Colorectal surgery

SUMMARY:
While perirenal fat measurement is an easy reproducible surrogate of visceral fat, its value as independent parameter in predicting postoperative complications after colorectal resection remains poorly investigated.

The investigators want to test the value of perirenal fat as surrogate of visceral obesity as risk factor for morbidity in colorectal surgery and to compare it to the effect of Body mass index (BMI) and Waist- Hip ratio (WHR).

ELIGIBILITY:
Inclusion Criteria:

* elective colorectal resection

Exclusion Criteria:

* age under 18
* emergency condition
* immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included all elective colorectal resections for benign, malignant and inflammatory diseases, admitted to the Geneva university hospital, Geneva, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  Postoperative complications (Clavien-Dindo classification)

SECONDARY OUTCOMES:
Duration of the operation | From incision to dressing of the wound
Rate of conversion | From incision to dressing of the wound

CONTACTS AND LOCATIONS:
Overall Officials: Minoa Jung, MD, Principal Investigator — University Hospital, Geneva; Francesco Volonte, MD, Principal Investigator — University Hospital, Geneva; Philippe Morel, MD, Study Chair — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland